CLINICAL TRIAL: NCT05886465
Title: Hepatic Arterial Infusion Chemotherapy With FOLFOX Plus Atezolizumab and Bevacizumab for Patients With High-risk Hepatocellular Carcinoma: a Single-arm Phase 2 Trial
Brief Title: HAIC Plus A+T for Patients With High-risk HCC: a Single-arm Phase 2 Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-014
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: High-risk hepatocellular Carcinoma; Hepatic arterial infusion chemotherapy; Oxaliplatin, 5-Fluorouracil and Leucovorin; Atezolizumab plus Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC plus A+T (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Procedure: HAIC with FOLFOX

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg, iv.drip, Q3W
Drug: Bevacizumab — 15mg/kg, iv.drip, Q3W
Procedure: HAIC with FOLFOX — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries, Q3W

SUMMARY:
Atezolizumab plus bevacizumab is the first-line treatment for patients with advanced hepatocellular carcinoma. However, the prognosis for high-risk hepatocellular carcinoma is still poor, with a median overall survival of 7.6 months. Hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin is effective in large hepatocellular carcinoma or hepatocellular carcinoma with major portal vein tumor thrombus. Our previous showed that hepatic arterial infusion chemotherapy plus lenvatinib and toripalimab (programmed cell death protein-1 antibody) had a powerful anti-tumor effect for high-risk hepatocellular carcinoma, with a median overall survival of 18 months. Thus, the purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin plus atezolizumab plus bevacizumab for patients with high-risk hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* High risk disease: Vp-4 based on the Japanese standard, bile duct invasion, or tumor occupancy ≥50% of the liver
* Eastern Cooperative Oncology Group performance status of 0 to 2
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate at 6 months | 6 months
  Progression was defined as progressive disease by independent radiologic review according to RECIST 1.1 or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS is the length of time from the date of randomization until death from any cause.
Progression free survival (PFS) | 6 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.
Adverse events | 30 days
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China